CLINICAL TRIAL: NCT03511391
Title: CHEckpoint Inhibition in Combination With an Immunoboost of External Beam Radiotherapy in Solid Tumors: CHEERS-trial
Brief Title: CHEckpoint Inhibition in Combination With an Immunoboost of External Beam Radiotherapy in Solid Tumors
Acronym: CHEERS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: GZA Ziekenhuizen Campus Sint-Augustinus (Other); AZ Sint-Lucas Brugge (Other); Jules Bordet Institute (Other); AZ Sint-Lucas Gent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC2017/1678
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Urothelial Carcinoma; Melanoma; Renal Cell Carcinoma; Non-small Cell Lung Cancer; Head and Neck Cancer
Keywords: radiotherapy; checkpoint inhibitors
MeSH Terms: conditions — Carcinoma, Transitional Cell; Melanoma; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms | interventions — Nivolumab; pembrolizumab; atezolizumab; Immune Checkpoint Inhibitors; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Stereotactic body radiotherapy concurrent with checkpoint inhibitor treatment:
  Nivolumab or Pembrolizumab or Atezolizumab + SBRT
  Interventions: Drug: Nivolumab or Pembrolizumab or Atezolizumab; Radiation: SBRT
- Control arm (Active Comparator): Checkpoint inhibitor treatment only:
  Nivolumab or Pembrolizumab or Atezolizumab monotherapy
  Interventions: Drug: Nivolumab or Pembrolizumab or Atezolizumab

INTERVENTIONS:
Drug: Nivolumab or Pembrolizumab or Atezolizumab — per national standard of care
  Other Names: Immune checkpoint inhibitor
Radiation: SBRT — Stereotactic body radiotherapy is administered to maximally 3 lesions in 3 fractions of 8Gy prior to the second/third cycle of checkpoint inhibitors.
  Other Names: Stereotactic body radiotherapy, SABR, Stereotactic ablative radiotherapy
  Arms: Experimental arm

SUMMARY:
This randomized controlled phase II trial will investigate whether the addition of stereotactic body radiotherapy to checkpoint inhibitor treatment in patients with non-small-cell lung carcinoma, urothelial carcinoma, renal cell carcinoma, melanoma or head-and-neck carcinoma can improve progression-free survival as compared to checkpoint inhibitor monotherapy. The primary outcome is progression-free survival; secondary outcomes include overall survival, response according to iRecist and Recist v1.1 and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Before patient registration, written informed consent must be given according to ICH/GCP and national/local regulations.
* Histologically confirmed diagnosis of a solid tumour.
* At least one extracranial tumour lesion available for radiotherapy administration.
* Patient will receive a checkpoint inhibitor per standard of care in one of the following settings (locally advanced or metastatic): melanoma (1st - 3rd line nivolumab or pembrolizumab); renal cell carcinoma (2nd line nivolumab); non-small cell lung carcinoma (2nd or 3rd line nivolumab, pembrolizumab or atezolizumab); urothelial cell carcinoma ( 1st-3rd line nivolumab, pembrolizumab or atezolizumab); head-& neck squamous cell carcinoma (1st-2nd line pembrolizumab, 2nd line nivolumab).
* Karnofsky Performance status > 60.
* Age 18 years or older.

Exclusion Criteria:

* Prior radiotherapy preventing treatment with SBRT.
* Prior treatment with an anti-PD-(L)1 antibody.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or prostate cancer that has undergone potentially curative therapy and with normalized PSA.
* Uncontrolled central nervous system (CNS) metastases at baseline (controlled = previously-treated CNS metastases (surgery ± radiotherapy, radiosurgery, or gamma knife) and who meet both of the following criteria: a) are asymptomatic and b) have no requirement for steroids or enzyme-inducing anticonvulsants), and/or carcinomatous meningitis.
* Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medication within 14 days prior to the first dose of study drug. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
* Has a diagnosis of immunodeficiency or history of human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C infection.
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study.
* Patient not likely to comply with the protocol; I.e. uncooperative attitude, inability to return for follow-up visits and unlikely to complete the study.
* Contraindication for radiotherapy.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 15 months
  Progression-free survival will be defined as the time from randomization to disease progression (as per iRECIST) or death from any cause.

SECONDARY OUTCOMES:
Overall survival | 2 years after start trial treatment
  Overall survival will be defined as the time from randomization to death from any cause.
Tumor response as per RECIST | 12 weeks
  Response of non-irradiated lesions will be evaluated as per RECIST v1.1.
Tumor response as per iRECIST | 12 weeks
  Response of non-irradiated lesions will be evaluated as per iRECIST
Incidence of Treatment-Related Adverse Events [safety and tolerability] | 12 weeks
  Adverse events will be monitored as per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Patient-reported quality of life | 12 weeks
  Quality of life will be assessed as per EORTC-QLQ C30 questionnaire
Systemic immune response | 12 weeks
  Exploratory translational analyses will be performed using blood and fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Piet Ost, PhD, Principal Investigator — University Ghent
Locations (5):
- Belgium (5):
  - AZ Sint-Lucas, Ghent, Oost-Vlaanderen
  - AZ Sint-Lucas, Bruges, West-Vlaanderen
  - GasthuisZusters Antwerpen, Antwerp
  - Jules Bordet Institute, Brussels
  - University Hospital Ghent, Ghent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Spaas M, Sundahl N, Kruse V, Rottey S, De Maeseneer D, Duprez F, Lievens Y, Surmont V, Brochez L, Reynders D, Danckaert W, Goetghebeur E, Van den Begin R, Van Gestel D, Renard V, Dirix P, Ost P. Checkpoint Inhibitors in Combination With Stereotactic Body Radiotherapy in Patients With Advanced Solid Tumors: The CHEERS Phase 2 Randomized Clinical Trial. JAMA Oncol. 2023 Sep 1;9(9):1205-1213. doi: 10.1001/jamaoncol.2023.2132. PMID 37410476
- [Derived] Spaas M, Sundahl N, Hulstaert E, Kruse V, Rottey S, De Maeseneer D, Surmont V, Meireson A, Brochez L, Reynders D, Goetghebeur E, Van den Begin R, Van Gestel D, Renard V, Dirix P, Mestdagh P, Ost P. Checkpoint inhibition in combination with an immunoboost of external beam radiotherapy in solid tumors (CHEERS): study protocol for a phase 2, open-label, randomized controlled trial. BMC Cancer. 2021 May 7;21(1):514. doi: 10.1186/s12885-021-08088-w. PMID 33962592